CLINICAL TRIAL: NCT06116045
Title: Phase 2 Clinical Study to Evaluate the Efficacy in Increasing Sexual Arousal, Safety and Tolerability of BZ371A in Gel Form Applied to Women with Sexual Arousal Disorder
Brief Title: Evaluation of the Efficacy, Safety and Tolerability of BZ371A in Women with Sexual Arousal Disorder
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Biozeus Biopharmaceutical S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BZ371CLI601
Record Dates: First submitted 2023-10-18; First posted 2023-11-03 (Actual); Last update posted 2024-10-22 (Actual); Status verified 2024-10

CONDITIONS: Female Sexual Arousal Disorder; Female Sexual Dysfunction
Keywords: Female; Sexual arousal disorder; Sexual dysfunction; FSFI questionnaire; Nitric Oxide; Topic
MeSH Terms: conditions — Sexual Dysfunctions, Psychological; Sexual Dysfunction, Physiological

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (6):
- Group A - BZ371A, then Placebo (Experimental): Participants will first receive topical BZ371A 7.5 mg for daily use for 2 weeks. After a washout period of 2 weeks, they will receive topical Placebo to be used daily for 2 weeks.
  Interventions: Drug: BZ371A 7.5 mg (1.5 ml); Drug: Placebo (1.5 ml)
- Group B - Placebo, then BZ371A (Experimental): Participants will first receive topical Placebo for daily use for 2 weeks. After a washout period of 2 weeks, they will receive topical BZ371A 7.5 mg to be used daily for 2 weeks.
  Interventions: Drug: BZ371A 7.5 mg (1.5 ml); Drug: Placebo (1.5 ml)
- Group C - BZ371A, then Placebo (Experimental): Participants will first receive topical BZ371A 5.0 mg for daily use for 2 weeks. After a washout period of 2 weeks, they will receive topical Placebo to be used daily for 2 weeks.
  Interventions: Drug: BZ371A 5.0 mg (1.0 ml); Drug: Placebo (1.0 ml)
- Gorup D - Placebo, then BZ371A (Experimental): Participants will first receive topical Placebo for daily use for 2 weeks. After a washout period of 2 weeks, they will receive topical BZ371A 5.0 mg to be used daily for 2 weeks.
  Interventions: Drug: BZ371A 5.0 mg (1.0 ml); Drug: Placebo (1.0 ml)
- Group E - BZ371A, then Placebo (Experimental): Participants will first receive topical BZ371A 2.5 mg for daily use for 2 weeks. After a washout period of 2 weeks, they will receive topical Placebo to be used daily for 2 weeks.
  Interventions: Drug: BZ371A 2.5 mg (0.5 ml); Drug: Placebo (0.5 ml)
- Group F - Placebo, then BZ371A (Experimental): Participants will first receive topical Placebo for daily use for 2 weeks. After a washout period of 2 weeks, they will receive topical BZ371A 2.5 mg to be used daily for 2 weeks.
  Interventions: Drug: BZ371A 2.5 mg (0.5 ml); Drug: Placebo (0.5 ml)

INTERVENTIONS:
Drug: BZ371A 7.5 mg (1.5 ml) — 7.5 mg gel
  Other Names: BZ371A
  Arms: Group A - BZ371A, then Placebo; Group B - Placebo, then BZ371A
Drug: BZ371A 5.0 mg (1.0 ml) — 5.0 mg gel
  Other Names: BZ371A
  Arms: Gorup D - Placebo, then BZ371A; Group C - BZ371A, then Placebo
Drug: BZ371A 2.5 mg (0.5 ml) — 2.5 mg gel
  Other Names: BZ371A
  Arms: Group E - BZ371A, then Placebo; Group F - Placebo, then BZ371A
Drug: Placebo (1.5 ml) — BZ371A-matched placebo
  Other Names: Placebo
  Arms: Group A - BZ371A, then Placebo; Group B - Placebo, then BZ371A
Drug: Placebo (1.0 ml) — BZ371A-matched placebo
  Other Names: Placebo
  Arms: Gorup D - Placebo, then BZ371A; Group C - BZ371A, then Placebo
Drug: Placebo (0.5 ml) — BZ371A-matched placebo
  Other Names: Placebo
  Arms: Group E - BZ371A, then Placebo; Group F - Placebo, then BZ371A

SUMMARY:
To determine the efficacy in increasing sexual arousal, safety and tolerability of BZ371A in gel form applied to women with sexual arousal disorder.

DETAILED DESCRIPTION:
FSAD is defined as the recurrent inability to attain or maintain sufficient genital arousal during sexual activity. Therefore, a healthy blood flow is central to the physiological processes related to sexual arousal, leading to genital lubrication, warmth, and clitoral protrusion.

The vasculature and blood flow in vaginal tissue can be compromised due to natural aging and various risk factors, including cigarette smoking, alcohol abuse, lack of exercise, high-fat diets, hypertension, hypercholesterolemia, and diabetes mellitus. All these risk factors and conditions are highly prevalent among women and can lead to FSAD. BZ371A offers a potential solution by increasing blood flow in genital tissue through its unique mechanism of action, thereby restoring vascular homeostasis and the physiological processes related to sexual arousal in women.

ELIGIBILITY:
Inclusion Criteria:

* Women between the ages 21 and 60;
* Pre-menopausal or post-menopausal women may be included;
* May or may not be taking female sex hormones (estrogen with or without progesterone, or their derivatives);
* FSAD, defined as the inability, persistent or recurrent, to obtain or maintain until the conclusion of sexual activity an adequate genital response to sexual arousal (lubrication, warmth and enlargement of the clitoris);
* Women with FSAD who present marked suffering or interpersonal difficulties;
* Stable relationship for more than 6 months, with a sexually active partner;
* Ability to read and understand the Informed Consent Form (ICF) and to answer the questionnaires.

Exclusion Criteria:

* Women who do not agree to use a contraceptive method and who have the capacity to become pregnant during the study;
* Women who do not agree to attempt sexual activity at least twice a week while taking the study medication;
* History of unresolved sexual trauma or abuse;
* Diagnosis of vaginismus, genitopelvic pain/penetration disorder and/or sexual aversion disorder;
* Uncontrolled diabetes at screening visit (HbA1C > 10%);
* Prior spinal cord injury, with lower limb paralysis;
* History of abdominal or pelvic surgery that may have damaged pelvic nerves, including vulvectomy, colostomy, cytostomy, hysterectomy, or bladder suspension.
* Current testosterone use, or long-term testosterone use (such as chip) within the past 6 months;
* Presence of menstrual irregularity or endocrinopathies that significantly alter the menstrual cycle, preventing Cytocam analyses from taking place at the same time;
* Patients with current depression, characterized by the use or need for use of psychotropic drugs, including bupropion, lithium, or neuroleptics;
* Presence of genital lesions that impair analysis of local adverse effects on the genitalia;
* Presence of diseases that cause excessive vaginal discharge, such as recurrent urinary tract infection, vaginal infection and pelvic inflammatory disease.
* Abnormal Papanicolaou test within the past 3 years;
* History of gynecological cancer (history of uterine dysplasia can be included, provided it has been properly treated for at least 6 months);
* History of pelvic irradiation;
* Use of topical medications in the genital region that may interfere with PSI assessment as well as their absorption or drug interaction, including vaginal estrogens, lubricants, spermicides, creams or gels, vaginal douches;
* History of symptomatic hypotension, or diseases that increase the risk of symptomatic hypotension, such as patient with heart disease (including history of angina and/or heart failure) and nephropathies;
* Current use of nitrates, such as propatylnitrate (Sustrate®), isosorbide (Monocordil®, Cincordil®, Isordil®), nitroglycerin (Nitradisc®, Nitroderm TTS®, Nitronal®, Tridil®) and sosorbitol dinitrate (Isocord®)
* ECG findings that are clinically symptomatic, or that, in the Investigator's judgment, are considered significant and pose a risk to the research volunteer's participation;
* Findings on laboratory tests that, in the Investigator's judgment, are considered significant and offer risk to the research volunteer's participation or may hinder the study analyses;
* TSH outside normal limits for age (participants with hypothyroidism on stable dose of medication, over 3 months, may be included);
* BP outside safe limits: SBP below 90 mmHg or above 170 mmHg; or DBP below 50 mmHg or above 100 mmHg, except for situations such as "white coat" syndrome
* Severe hypertension, considered as use of three or more antihypertensives;
* Diseases that can cause clitoral priapism, such as sickle cell anemia, multiple myeloma or leukemia;
* History of clitoral priapism;
* Current relevant diarrhea, defined as duration over four weeks, association with abdominal pain or malabsorptive syndrome, or presence of mucus, pus, or blood in the stool;
* Pregnant or lactating;
* Current use of nitric oxide donors, guanylate cyclase stimulators (e.g. Riociguat), or 5- phosphodiesterase inhibitors (Sildenafil, Tadalafil, etc.);
* Any disease or condition or physical finding that the Investigator considers significant and that increases the risk of the research participant's participation or may interfere with the results, including serious debilitating diseases, presence of cancer, serious mental illness, persistent abuse of medication.

Ages: 21 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-03-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy in increasing arousal | Baseline, 4 weeks and 8 weeks
  Evaluation of the efficacy of BZ371A in increasing arousal using Female Sexual Encounter Profile (FSEP) questionnaire. The study will evaluate number of "yes" answers to question 3 in the Female Sexual Encounter Profile (FSEP) questionnaire, divided by the number of valid attempts (question 7 of the FSEP).
  The study will evaluate the increase in the FSEP score based on the baseline FSEP value, obtained before using the BZ371A. Thus, the higher the number of yes answers, the better the efficacy of the drug.

SECONDARY OUTCOMES:
Efficacy in increasing desire, lubrification, orgasm and arousal | Baseline, 4 weeks and 8 weeks
  Evaluation of the success rate for desire, lubrification, orgasm and for arousal using Female Sexual Encounter Profile (FSEP). The number of successes for desire will be assessed using FSEP Question 2 / FSEP Question 7, for lubrication FSEP Question 4 / FSEP Question 7, for orgasm FSEP Question 5 / FSEP Question 7 and for the degree of arousal FSEP Question 6 / FSEP Question 7.
  For each question, the number of "yes" answers will be counted as success. Therefore, for each "no" answer the value will be 0 and for each "yes" answer the value will be 1.
Evaluation of the quality of female sexual encounters | Baseline, 4 weeks and 8 weeks
  Evaluation based on the total score of the Female Sexual Encounter Profile (FSEP) questionnaire. The score ranges from 0 to 9. Therefore, the higher the score, the better the participant's sexual encounter.
Efficacy in increasing genital blood flow | Baseline, 4 weeks (pre-dose, 15, 30, 60, 90 and 120 minutes) and 8 weeks (pre-dose, 15, 30, 60, 90 and120 minutes)
  Evaluation of the efficacy of BZ371A in increasing genital blood flow using Cytocam system
Female Sexual Function Index (FSFI) | Baseline, 4 weeks and 8 weeks
  Evaluation of the score for each domain (Desire, Arousal, Lubrication, Orgasm, Satisfaction, Pain) using the Female Sexual Function Index (FSFI) questionnaire. The score ranges from 2 to 36. Thus, the higher the score, the better the participant's sexual satisfaction.
Assessment of treatment satisfaction | 4 weeks after baseline and 8 weeks after baseline
  Response rate to the Global Assessment Question (GAQ), by the number of "yes" answers to the question about arousal and sexual pleasure.
Adverse effects report | 4 weeks after baseline, 8 weeks after baseline and, approximately, 11 weeks after baseline
  Adverse effects evaluation of compound use and application
Physical examination of the genitalia | From up to 30 days before Baseline, Baseline, 4 weeks, 8 weeks and, approximately, 11 weeks
  Number of participants with abnormal physical exam findings in the applied region.
Change in systemic blood pressure | From up to 30 days before Baseline, Baseline, 4 weeks, 8 weeks and, approximately, 11 weeks
  Change in Diastolic Blood Pressure and Systolic Blood Pressure
Change in Heart Rate (HR) | From up to 30 days before Baseline, Baseline, 4 weeks, 8 weeks and, approximately, 11 weeks
  Change in Heart Rate
Basal chest electrocardiogram (ECG) | From up to 30 days before Baseline, 4 weeks after baseline, 8 weeks after baseline
  Number of participants with abnormal electrocardiogram (ECG) findings.
Blood evaluation | From up to 30 days before Baseline, 4 weeks after baseline and 8 weeks after baseline
  Number of participants with abnormal laboratory test results
Urine evaluation | From up to 30 days before Baseline, 4 weeks after baseline and 8 weeks after baseline
  Number of participants with abnormal laboratory test results

CONTACTS AND LOCATIONS:
Overall Officials: Marco Aurélio Oliveira, MD, Principal Investigator — Centro de Pesquisa Clínica Multiusuário (CePeM)
Locations (1):
- Centro de Pesquisa Clínica Multiusuário (CePeM), Rio de Janeiro, Rio de Janeiro, Brazil